CLINICAL TRIAL: NCT03252821
Title: Effects of High-intensity Training Compared to Resistance Training in Cancer Patients Undergoing Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Caty Gilles, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-07-31; First posted 2017-08-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer; Head and Neck Cancer; Rectum Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Head and Neck Neoplasms; Rectal Neoplasms | interventions — High-Intensity Interval Training; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity aerobic training group (Experimental): High intensity interval training
  Interventions: Behavioral: High-intensity interval training
- Resistance training group (Active Comparator): Muscle strengthening
  Interventions: Behavioral: Resistance training
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: High-intensity interval training — High-intensity interval training sessions will be conducted on cycle ergometers or treadmill with heart rate measured throughout each session.
  Arms: High-intensity aerobic training group
Behavioral: Resistance training — Resistance exercise will be performed on eight exercises targeting major muscle groups at 60% to 85% of their estimated one-repetition maximum (1RM).
  Arms: Resistance training group

SUMMARY:
The aim of this study is to assess the impact of a high-intensity aerobic training and resistance training on fatigue in prostate, head and neck and rectum cancer patients undergoing radiotherapy.

A three-arm randomized controlled trial will be conducted. Patients will be randomised into either a high-intensity aerobic training group or a resistance training group or a control group. Participants in the training groups will exercised for five to eight weeks. Exercise sessions will be take place 3 days per week under the supervision of an experienced therapist. Subjects will be assessed at baseline and post-intervention. The primary outcome will be fatigue measured using the FACIT-fatigue questionnaire. The secondary outcomes will be: functional capacity, quality of life, executive functions, sleep disturbances, somnolence syndrome, insomnia, depression symptoms.

ELIGIBILITY:
Inclusion criteria :

* a primary diagnosis of prostate cancer, head and neck cancer (oral cavity, pharynx, larynx, nasal cavity/sinuses, or salivary gland) or rectum cancer;
* age over 18 years;
* no distant metastases and/or disease progression;
* at least 25 scheduled radiation treatments (5 weeks);
* ability to read, write, and speak French.

Exclusion criteria :

* uncontrolled cardiac, hypertensive or pulmonary diseases,
* uncontrolled insulin-dependent diabetes mellitus,
* neuropsychiatric disorders or orthopaedic conditions that would impair exercise participation
* abnormal electrocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Change in fatigue | Assessments at baseline and 5 weeks (rectum cancer) or 7 weeks (head and neck cancer) or 8 weeks (prostate cancer)
  Fatigue is measured by FACIT-fatigue questionnaire

SECONDARY OUTCOMES:
Change in functional capacity | Assessments at baseline and 5 weeks (rectum cancer) or 7 weeks (head and neck cancer) or 8 weeks (prostate cancer)
  Functional capacity is measured by 6-minute walk test
Change in quality of life | Assessments at baseline and 5 weeks (rectum cancer) or 7 weeks (head and neck cancer) or 8 weeks (prostate cancer)
  Quality of life is measured by Functional Assessment of Cancer Therapy-General
Change in sleep disturbances | Assessments at baseline and 5 weeks (rectum cancer) or 7 weeks (head and neck cancer) or 8 weeks (prostate cancer)
  Sleep disturbances are measured by Pittsburgh Sleep Quality Index
Change in somnolence syndrome | Assessments at baseline and 5 weeks (rectum cancer) or 7 weeks (head and neck cancer) or 8 weeks (prostate cancer)
  Somnolence syndrome is measured by Epworth Sleepiness Scale
Change in insomnia | Assessments at baseline and 5 weeks (rectum cancer) or 7 weeks (head and neck cancer) or 8 weeks (prostate cancer)
  Insomnia is measured by Insomnia Severity Index
Change in depression symptoms | Assessments at baseline and 5 weeks (rectum cancer) or 7 weeks (head and neck cancer) or 8 weeks (prostate cancer)
  Depression symptoms are measured by Center for Epidemiologic Studies Depression Scale
Change in executive functions | Assessments at baseline and 5 weeks (rectum cancer) or 7 weeks (head and neck cancer) or 8 weeks (prostate cancer)
  Executive functions is measured by the Trail Making Test
Change in dyspnea | Assessments at baseline and 5 weeks (rectum cancer) or 7 weeks (head and neck cancer) or 8 weeks (prostate cancer)
  Dyspnea is measured by Multidimensional Dyspnea Profile
Adherence | Weekly through the intervention (during 8 weeks)
  Percentage of completed sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Piraux E, Reychler G, Vancraeynest D, Geets X, Leonard D, Caty G. High-intensity aerobic interval training and resistance training are feasible in rectal cancer patients undergoing chemoradiotherapy: a feasibility randomized controlled study. Rep Pract Oncol Radiother. 2022 May 19;27(2):198-208. doi: 10.5603/RPOR.a2022.0036. eCollection 2022. PMID 36299392